CLINICAL TRIAL: NCT06160076
Title: Inflammatory Response Following " Pulsed Field Ablation " vs. Radiofrequency Ablation of Paroxysmal Atrial Fibrillation-2
Brief Title: Inflammatory Response Following " Pulsed Field Ablation " vs. Radiofrequency Ablation-2
Acronym: RIPAF-2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2023/33
Record Dates: First submitted 2023-09-28; First posted 2023-12-07 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Atrial Fibrillation; Catheter Ablation; Inflammation
Keywords: Atrial Fibrillation; catheter ablation; Inflammation; Pulsed-field ablation
MeSH Terms: conditions — Atrial Fibrillation; Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Radiofrequency: Patient with atrial fibrillation ablated per radiofrequency
  Interventions: Device: Radiofrequency
- Pulsed electric field: Patient with atrial fibrillation ablated per pulsed electric field
  Interventions: Device: Pulsed electric field

INTERVENTIONS:
Device: Radiofrequency — Patient with atrial fibrillation ablated per catheter using radiofrequency energy
  Other Names: Catheter ablation per radiofrequency
  Groups: Radiofrequency
Device: Pulsed electric field — Patient with atrial fibrillation ablated per catheter using pulsed electric field
  Other Names: Catheter ablation per pulsed electric field
  Groups: Pulsed electric field

SUMMARY:
Atrial fibrillation (AF) is the most common sustained cardiac arrhythmia. Catheter ablation using pulmonary vein isolation (PVI) in an established treatment strategy for AF. Pulsed Field Ablation (PFA) is a non-thermal ablation modality which has recently been introduced in clinical practice with the aim of improving PVI efficacy and safety. The aim of this study is to analyse whether PFA generates a lower inflammatory reaction as compared to conventional radiofrequency ablation (RFA).

DETAILED DESCRIPTION:
Pulmonary vein isolation represents the cornerstone of AF ablation. PFA is a novel non-thermal cardiac ablation modality which is currently studied in clinical trials for the treatment of AF with promising efficacy and safety results. PFA is reported to generate less collateral damage by inducing selective apoptosis of cardiomyocytes, while other structures such as nerves, vessels and oesophageal tissue remain spared. PFA lesions show more organized and homogeneous fibrosis on histopathological study as compared to thermal lesions. In a recent study conducted at Hôpital Haut-Lévêque, PFA was associated with 20% less acute oedema on magnetic resonance imaging. Therefore, PFA may generate a reduced inflammatory reaction which could translate into lower early recurrence rates, less post-procedural chest pain and improved clinical outcomes. Data on the systemic inflammation generated by PFA and RFA is still lacking.

The aim of this study is to analyse the inflammatory reaction after PFA and RFA in patients referred for first-time catheter ablation of paroxysmal AF. For this purpose, established biomarkers of systemic inflammation (leucocytosis, platelet-monocyte-complexes, inflammatory cytokines) will be determined in blood samples collected from patients treated with either PFA or RFA.

The collection of blood samples will be exclusively performed during routine blood drawing at three time points: at the beginning of the procedure (to define baseline values), at the end of the procedure (to measure acute inflammation) and the day following the procedure (to define inflammation occurring within 24 hours). Clinical signs of inflammation (fever, chest pain, pericardial fluid) and early arrhythmia recurrences will also be assessed the day after the ablation. On a routine 6-month follow-up visit, late arrhythmia recurrences will be registered. In a secondary analysis, the thrombogenic and pro-arrhythmogenic potential of both ablation modalities and the predictive value of inflammatory biomarkers for early and late recurrences will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with paroxysmal AF referred for first-time catheter ablation using PFA or RFA
* Non-opposition to participate

Exclusion Criteria:

* Age < 18 years
* Persons under judicial protection (guardianship, guardianship) or deprived of freedom
* Prior left atrial ablation
* Prior cardiac surgery comprising incision of the left atrium
* Prior myocardial infarction or stroke in the previous 30 days
* Acute or chronic inflammatory state: active smoking, auto-immune disease, active tumor disease, myocarditis
* Antiplatelet therapy (e.g. aspirine, clopidogrel) within the 7 last days
* Anti-inflammatory treatment (e.g. glucocorticoids, colchicine, cyclophosphamide, azathioprine, mycophenolic acid, antibodies) within the 7 last days

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation treated by catheter ablation
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
Acute thromboinflammatory response | 24 hours
  Circulating platelet-monocyte complexes (PMC)
Systemic inflammatory response (IL-6) | 24 hours
  Changes in leukocyte count and circulating levels of IL-6
Systemic inflammatory response (TNF-α) | 24 hours
  Changes in leukocyte count and circulating levels of TNF-α
Systemic inflammatory response (CRP) | 24 hours
  Changes in leukocyte count and circulating levels of CRP
Pericarditis | 24 hours
  Chest pain suggestive of pericarditis assessed using a numeric pain rating scale (0 to 10)

SECONDARY OUTCOMES:
Incidence of early arrhythmias | 24 hours
  Incidence of early arrhythmias occurring during the post-operative period on telemetry in PFA vs. RFA
Analysis of biomarkers (CD40L) | 24 hours
  Platelet activation: Changes in plasma levels of soluble CD40L
Analysis of biomarkers (Willebrand) | 24 hours
  Endothelial cell damage: Changes in plasma levels of von Willebrand factor
Incidence of late atrial arrhythmia recurrence | 6 months
  Atrial fibrillation and/or atrial tachycardia recurrences documented by Holter-ECGs or other wearable devices

CONTACTS AND LOCATIONS:
Overall Officials: Pierre JAÏS, MD, Study Director — University Hospital, Bordeaux
Locations (1):
- Hôpital Haut-Lévèque, Pessac, France

IPD SHARING:
Plan to Share IPD: No